CLINICAL TRIAL: NCT03996642
Title: Feasibility of Delivering an Avatar Life-review Intervention to Support Patients With Active Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Massey Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: MCC-18-14462; HM20014524 (Other: IRB); MCC-18-14462: (Other Grant/Funding Number: Massey Cancer Center); NCI-2019-03865 (Other: NCI)
Record Dates: First submitted 2019-06-11; First posted 2019-06-25 (Actual); Last update posted 2020-02-06 (Actual); Status verified 2020-02

CONDITIONS: Cancer
Keywords: active; cancer; avatar; life-limiting; palliative care
MeSH Terms: conditions — Neoplasms; Motor Activity

STUDY DESIGN:
Intervention Model Description: This study will use a one-group observational design to establish feasibility and acceptability of Avatar therapy intervention in patients with advanced cancer.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with Active Cancer (Other): Eligible participants will undergo an unknown number of Avatar-life review sessions depending on acceptability of the intervention to subjects and the capacity of the team to provide the intervention.
  Interventions: Behavioral: Avatar Life Review

INTERVENTIONS:
Behavioral: Avatar Life Review — VoicingHan will screen-capture patient's storytelling performances as video files. Immediately before the first intervention, patients will complete an array of self-reported questionnaires to assess physical, spiritual, and psychological well-being and elicit relevant demographic and medical information. The assessments include the ESAS, FACIT-Sp subscale, and EORTC PAL 15. Subsequent administration of these questionnaires spaced 2-4 weeks apart will occur before each avatar session (pre-intervention). This will determine if intensity of the patient's symptoms have changed over the course of the intervention. Following completion of the Avatar session, a member of the research team will conduct a semi-structured, open-ended interview to assess patients' perception of intervention components and identify possible factors influencing intervention feasibility and any technical barriers.

SUMMARY:
The objective of the study is to determine the feasibility and acceptability of an integrated art and technology, storytelling, life review platform for patients with active cancer. The VoicingHan project is an avatar storytelling platform designed for patients with advanced cancer receiving palliative care at Virginia Commonwealth University's Massey Cancer Center. VoicingHan supports terminally ill patients by using oral storytelling as an artistic medium to facilitate patients' interactive performances. Movement-based, creative expression has been shown to reduce stress and depression. By projecting movement-based actions onto an avatar, this can serve as a tool to express emotional distress, address satisfaction with care, and view cancer in a different light.

DETAILED DESCRIPTION:
Life reviews have been used in palliative care to help individuals integrate memories into a meaningful whole, providing a balanced view of the past, present and future. Life review is also an evaluative process, enabling participants to examine how memories contribute to the meaning of their life.

VoicingHan, the software program that will be used in this study, provides an illusion that the Avatar is speaking, allowing users to observe their stories in real time, potentially encouraging deeper reflection and memory retrieval. The technology uses motion capture (MoCap) to translate human movement into a digital platform. MoCap offers several advantages: lightweight, sensitive to minute movement, and user-friendly.

Patients will select avatars from different age groups during their sessions, allowing them to retrieve specific, positive memories of different lifetime periods and facilitating a more candid autobiographical memory. Creative expression may serve as a vehicle for patients with a life limiting illness in finding purpose and creating a sense of meaning. The integration of art and technology into a storytelling, life-review platform through means of engaging the physical, psychological, and spiritual domains will support patients to contemplate their own mortality.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be 18 years of age or older
* Patient participants must have metastatic or locally recurrent cancer
* Participants must be able to understand English
* Participants must be ambulatory
* Ability and willingness to sign a written informed consent document

Exclusion Criteria:

* Participants who cannot understand written or spoken English
* Any prisoner and/or other vulnerable persons as defined by NIH (45 CFR 46, Subpart B, C and D).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2019-07-19 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-10-23 (Actual)

PRIMARY OUTCOMES:
Portion of successfully completed sessions | 2 months
  The total number of sessions completed in compliance with the required protocol divided by the total number of sessions attempted
Patient's perceived benefits of intervention | 15 minutes
  The research coordinator will conduct an open-ended interview to assess patients' perception of intervention components and identify possible factors influencing feasibility. Questions will address feasibility of setup time, study procedure, and level of comfort
The ability to recruit patients to participate in the Avatar Therapy intervention | 2 months
  Feasibility of recruitment efforts will be determined by the proportion of patients that are enrolled divided by the number of patients contacted and approached to participate.

SECONDARY OUTCOMES:
Determine length of time required to set-up the technology | 10 minutes
  length of setup time as determined when first entering the outpatient room to the arrival of the patient
Determine the average time per session for each participant | 60 minutes
  Length of session as determined by the start of participant's arrival to their departure.
Determine the number of intervention sessions needed per patient | 5 minutes
  Participants will complete a 3 item brief survey administered by the research coordinator at the end of each session to determine if patients would benefit from another avatar session. Each item is rated on a five-point Likert scale from "1= Not at all to "5= A lot/Extremely" with higher scores indicating greater patient satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Egidio Del Fabbro, MD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Coelho A, Parola V, Cardoso D, Bravo ME, Apostolo J. Use of non-pharmacological interventions for comforting patients in palliative care: a scoping review. JBI Database System Rev Implement Rep. 2017 Jul;15(7):1867-1904. doi: 10.11124/JBISRIR-2016-003204. PMID 28708751
- [Background] Zabora J, BrintzenhofeSzoc K, Curbow B, Hooker C, Piantadosi S. The prevalence of psychological distress by cancer site. Psychooncology. 2001 Jan-Feb;10(1):19-28. doi: 10.1002/1099-1611(200101/02)10:13.0.co;2-6. PMID 11180574
- [Background] Lopez G, Garcia MK, Liu W, Spano M, Underwood S, Dibaj SS, Li Y, Moguel R, Williams J, Bruera E, Cohen L. Outpatient acupuncture effects on patient self-reported symptoms in oncology care: a retrospective analysis. J Cancer. 2018 Sep 8;9(19):3613-3619. doi: 10.7150/jca.26527. eCollection 2018. PMID 30310519
- [Background] Del Fabbro E, Dalal S, Bruera E. Symptom control in palliative care--Part III: dyspnea and delirium. J Palliat Med. 2006 Apr;9(2):422-36. doi: 10.1089/jpm.2006.9.422. No abstract available. PMID 16629572
- [Background] Singer AE, Goebel JR, Kim YS, Dy SM, Ahluwalia SC, Clifford M, Dzeng E, O'Hanlon CE, Motala A, Walling AM, Goldberg J, Meeker D, Ochotorena C, Shanman R, Cui M, Lorenz KA. Populations and Interventions for Palliative and End-of-Life Care: A Systematic Review. J Palliat Med. 2016 Sep;19(9):995-1008. doi: 10.1089/jpm.2015.0367. Epub 2016 Aug 17. PMID 27533892
- [Background] Holland J, Poppito S, Nelson C, Weiss T, Greenstein M, Martin A, Thirakul P, Roth A. Reappraisal in the eighth life cycle stage: a theoretical psychoeducational intervention in elderly patients with cancer. Palliat Support Care. 2009 Sep;7(3):271-9. doi: 10.1017/S1478951509990198. PMID 19788768
- [Background] Ryu S, Imaging K, Commonwealth V, Society K. Avatar life-review : Virtual bodies in a dramatic paradox. 2017;7(2):5-8. doi:10.1386/vcr.7.2.121
- [Background] World Health Organization. National Cancer Control Programmes. Natl cancer Control Program Policies Manag Guid. 2002:180. http://www.hdnet.org.
- [Background] Rhondali W, Lasserre E, Filbet M. Art therapy among palliative care inpatients with advanced cancer. Palliat Med. 2013 Jun;27(6):571-2. doi: 10.1177/0269216312471413. No abstract available. PMID 23685771
- [Background] Wood MJ, Molassiotis A, Payne S. What research evidence is there for the use of art therapy in the management of symptoms in adults with cancer? A systematic review. Psychooncology. 2011 Feb;20(2):135-45. doi: 10.1002/pon.1722. PMID 20878827
- [Background] Haber D. Life review: implementation, theory, research, and therapy. Int J Aging Hum Dev. 2006;63(2):153-71. doi: 10.2190/DA9G-RHK5-N9JP-T6CC. PMID 17137032
- [Background] van der Spek N, Vos J, van Uden-Kraan CF, Breitbart W, Cuijpers P, Holtmaat K, Witte BI, Tollenaar RAEM, Verdonck-de Leeuw IM. Efficacy of meaning-centered group psychotherapy for cancer survivors: a randomized controlled trial. Psychol Med. 2017 Aug;47(11):1990-2001. doi: 10.1017/S0033291717000447. Epub 2017 Apr 4. PMID 28374663
- [Background] Chochinov HM, Kristjanson LJ, Breitbart W, McClement S, Hack TF, Hassard T, Harlos M. Effect of dignity therapy on distress and end-of-life experience in terminally ill patients: a randomised controlled trial. Lancet Oncol. 2011 Aug;12(8):753-62. doi: 10.1016/S1470-2045(11)70153-X. Epub 2011 Jul 6. PMID 21741309
- [Background] Breitbart W, Poppito S, Rosenfeld B, Vickers AJ, Li Y, Abbey J, Olden M, Pessin H, Lichtenthal W, Sjoberg D, Cassileth BR. Pilot randomized controlled trial of individual meaning-centered psychotherapy for patients with advanced cancer. J Clin Oncol. 2012 Apr 20;30(12):1304-9. doi: 10.1200/JCO.2011.36.2517. Epub 2012 Feb 27. PMID 22370330
- [Background] Kleijn G, Lissenberg-Witte BI, Bohlmeijer ET, Steunenberg B, Knipscheer-Kuijpers K, Willemsen V, Becker A, Smit EF, Eeltink CM, Bruynzeel AME, van der Vorst M, de Bree R, Leemans CR, van den Brekel MWM, Cuijpers P, Verdonck-de Leeuw IM. The efficacy of Life Review Therapy combined with Memory Specificity Training (LRT-MST) targeting cancer patients in palliative care: A randomized controlled trial. PLoS One. 2018 May 15;13(5):e0197277. doi: 10.1371/journal.pone.0197277. eCollection 2018. PMID 29763431
- [Background] Xiao H, Kwong E, Pang S, Mok E. Effect of a life review program for Chinese patients with advanced cancer: a randomized controlled trial. Cancer Nurs. 2013 Jul-Aug;36(4):274-83. doi: 10.1097/NCC.0b013e318268f7ba. PMID 23047792
- [Background] Ando M, Morita T, Akechi T, Okamoto T; Japanese Task Force for Spiritual Care. Efficacy of short-term life-review interviews on the spiritual well-being of terminally ill cancer patients. J Pain Symptom Manage. 2010 Jun;39(6):993-1002. doi: 10.1016/j.jpainsymman.2009.11.320. PMID 20538183
- [Background] Gordon MS, Carswell SB, Schadegg M, Mangen K, Merkel K, Tangires S, Vocci FJ. Avatar-assisted therapy: a proof-of-concept pilot study of a novel technology-based intervention to treat substance use disorders. Am J Drug Alcohol Abuse. 2017 Sep;43(5):518-524. doi: 10.1080/00952990.2017.1280816. Epub 2017 Feb 17. PMID 28635345
- [Background] Craig TK, Rus-Calafell M, Ward T, Leff JP, Huckvale M, Howarth E, Emsley R, Garety PA. AVATAR therapy for auditory verbal hallucinations in people with psychosis: a single-blind, randomised controlled trial. Lancet Psychiatry. 2018 Jan;5(1):31-40. doi: 10.1016/S2215-0366(17)30427-3. Epub 2017 Nov 23. PMID 29175276
- [Background] Stuckey HL, Nobel J. The connection between art, healing, and public health: a review of current literature. Am J Public Health. 2010 Feb;100(2):254-63. doi: 10.2105/AJPH.2008.156497. Epub 2009 Dec 17. PMID 20019311
- [Background] Bruera E, Kuehn N, Miller MJ, Selmser P, Macmillan K. The Edmonton Symptom Assessment System (ESAS): a simple method for the assessment of palliative care patients. J Palliat Care. 1991 Summer;7(2):6-9. PMID 1714502
- [Background] Chang VT, Hwang SS, Feuerman M. Validation of the Edmonton Symptom Assessment Scale. Cancer. 2000 May 1;88(9):2164-71. doi: 10.1002/(sici)1097-0142(20000501)88:93.0.co;2-5. PMID 10813730
- [Background] Groenvold M, Klee MC, Sprangers MA, Aaronson NK. Validation of the EORTC QLQ-C30 quality of life questionnaire through combined qualitative and quantitative assessment of patient-observer agreement. J Clin Epidemiol. 1997 Apr;50(4):441-50. doi: 10.1016/s0895-4356(96)00428-3. PMID 9179103
- [Background] Breitbart W, Rosenfeld B, Gibson C, Pessin H, Poppito S, Nelson C, Tomarken A, Timm AK, Berg A, Jacobson C, Sorger B, Abbey J, Olden M. Meaning-centered group psychotherapy for patients with advanced cancer: a pilot randomized controlled trial. Psychooncology. 2010 Jan;19(1):21-8. doi: 10.1002/pon.1556. PMID 19274623
- [Background] van Belle G. Statistical Rules of Thumb. New York : John Wiley and Sons, 2002
- [Background] Julious, S. A. (2005), Sample size of 12 per group rule of thumb for a pilot study. Pharmaceut. Statist., 4: 287-291. doi:10.1002/pst.185
- [Result] Brady MJ, Peterman AH, Fitchett G, Mo M, Cella D. A case for including spirituality in quality of life measurement in oncology. Psychooncology. 1999 Sep-Oct;8(5):417-28. doi: 10.1002/(sici)1099-1611(199909/10)8:53.0.co;2-4. PMID 10559801
- [Derived] Dang M, Noreika D, Ryu S, Sima A, Ashton H, Ondris B, Coley F, Nestler J, Fabbro ED. Feasibility of Delivering an Avatar-Facilitated Life Review Intervention for Patients with Cancer. J Palliat Med. 2021 Apr;24(4):520-526. doi: 10.1089/jpm.2020.0020. Epub 2020 Sep 3. PMID 32896200

DOCUMENTS (1):
  • Informed Consent Form (2019-05-31): https://cdn.clinicaltrials.gov/large-docs/42/NCT03996642/ICF_002.pdf